CLINICAL TRIAL: NCT05277948
Title: Effect of Thumbtack Needle on Ovarian Function of Women With Diminished Ovarian Reserve (DOR): A Randomized Controlled Clinical Trial
Brief Title: Effect of Thumbtack Needle on Ovarian Function of Women With Diminished Ovarian Reserve (DOR)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Dongmei Huang, associate Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Effect of TTN on DOR
Record Dates: First submitted 2021-12-22; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Diminished Ovarian Reserve

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Active Comparator): Active thumbtack needle will be used for the treatment group
  Interventions: Other: active thumbtack needle
- control group (Sham Comparator): Sham thumbtack needle will be used for the control group
  Interventions: Other: sham thumbtack needle

INTERVENTIONS:
Other: active thumbtack needle — The following 12 acupoints including conception vessel (CV) 4, CV3, bilateral ovary acupoints, bilateral spleen (SP) 6, bilateral stomach (ST) 36, bilateral bladder (BL) 23 and bilateral EX-B7 will be used. Eight points of CV4, CV3, SP6, ST36 and BL23 were treated by the sterile thumbtack needle for single use (Hangzhou Zhuomai Medical Technology Co., LTD., model: ZM2-6YDL), and four points of bilateral ovary acupoints and bilateral EX-B7 were treated by disposable sterile electro-thumbtack needle (Hangzhou Zhuomai Medical Technology Co., LTD., model: ZM3-ZY).
  The patients were receive a treatment of 2 menstrual cycles
  Arms: treatment group
Other: sham thumbtack needle — The following 12 acupoints including conception vessel (CV) 4, CV3, bilateral ovary acupoints, bilateral spleen (SP) 6, bilateral stomach (ST) 36, bilateral bladder (BL) 23 and bilateral EX-B7 will be used. Eight points of CV4, CV3, SP6, ST36 and BL23 were treated by the sterile sham thumbtack needle for single use (Hangzhou Zhuomai Medical Technology Co., LTD., model: ZM2-6YDL), and four points of bilateral ovary acupoints and bilateral EX-B7 were treated by disposable sterile sham electro-thumbtack needle (Hangzhou Zhuomai Medical Technology Co., LTD., model: ZM3-ZY).
  The patients were receive a treatment of 2 menstrual cycles
  Arms: control group

SUMMARY:
Using a multi-center, large sample, randomized, controlled and blind clinical trial to evaluate the effect of thumbtack needle on ovarian function of patients with diminished ovarian reserve (DOR).

DETAILED DESCRIPTION:
Diminished ovarian reserve (DOR) is the precursor state of ovarian failure, and can cause the decline of women's reproductive function. Some studies have demonstrated that acupuncture can improve ovarian function. Thumbtack needle, as a kind of acupuncture, has been found effective in treating DOR in our clinic. In this trial, the investigators Using a multi-center, large sample, randomized, controlled and blind clinical trial to evaluate the effect of thumbtack needle on ovarian function of patients with diminished ovarian reserve (DOR).

First, patients will be recruited according to the inclusion criteria and exclusion criteria.

Second, baseline measurements (including ovarian reserve function, blood biochemical index, scores from the self-rating anxiety and depression scale, quality of life, sleep status) will be taken.

Third, each patient will receive the treatment of thumbtack needle for a total of 2 menstrual cycles.

Last, the above baseline measurements will be taken again as soon as the treatment is finished and outcome measures will be recorded after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18 and 40 years;
* Low ovarian reserve: AMH<1.1ng/ml; or AFC<7; or 10 U/L<FSH<25U/L or FSH/LH>3.6; or has a history of poor ovarian response, that is, in the last controlled hyperstimulation cycle, the number of retrieved oocytes<3. Any 2 of the above 4 conditions are met.
* Sign informed consent voluntarily.

Exclusion Criteria:

* Patient's chromosome is abnormal.
* Patients with previous ovarian surgery because of such as ovarian teratoma or chocolate cyst and so on.
* Patients with uncorrected endocrine disease, such as: Simple hyperthyroidism or hypothyroidism, hyperprolactinemia, insulin resistance, diabetes, adrenal diseases, etc.
* Patients with definitively diagnosed autoimmune diseases such as systemic lupus erythematosus, rheumatoid arthritis, antiphospholipid syndrome, Sjogren's syndrome, Hashimoto's thyroiditis.
* Patients with a history of cancer and has received radiotherapy or chemotherapy.
* Patients had the treatment of acupuncture or thumbtack needle in recent 3 months.
* Patients who take Chinese medicine decoction or granule during the treatment;
* Patients unwilling to sign the informed consent of this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluating the change of serum AMH level | 0 week and up to 4 weeks
  Assessing patients' serum level of AMH in ng/ml at baseline and immediately after treatment on the second day of menstruation.
Evaluating the change of the ovarian antral follicle count (AFC) | 0 week and up to 4 weeks
  Counting the number of ovarian antral follicle count (AFC) on the second day of menstruation at baseline and immediately after treatment.

SECONDARY OUTCOMES:
Evaluating the serum levels of sex hormones | 0 week and up to 4 weeks
  Evaluating the serum levels of sex hormones on the second day of menstruation at baseline and immediately after treatment
Observing the sex hormones in follicular fluid collected from patients undergoing IVF/ICSI-ET cycle after treatment | through study completion, an average of 1 year
  Observing follicular fluid levels of sex hormones when patients undergoing IVF/ICSI
  -ET after the treatment.
Observing the level of transforming growth factor β (TGF β) in follicular fluid | through study completion, an average of 1 year
  Observing follicular fluid level of transforming growth factor β (TGF β) when patients undergoing IVF/ICSI
  -ET after the treatment.
Observing the level of tumor necrosis factor-α (TNF-α) in follicular fluid | through study completion, an average of 1 year
  Observing follicular fluid level of TNF-α when patients undergoing IVF/ICSI
  -ET after the treatment.
Observing the level of reactive oxygen species (ROS) in follicular fluid | through study completion, an average of 1 year
  Observing follicular fluid level of ROS when patients undergoing IVF/ICSI
  -ET after the treatment.
Observing the level of superoxide dismutase (SOD) in follicular fluid | through study completion, an average of 1 year
  Observing follicular fluid level of SOD when patients undergoing IVF/ICSI
  -ET after the treatment.
Observing the ovum morphology (MII ovum ratio) during IVF-ET after treatment | through study completion, an average of 1 year
  Observing the MII ovum ratio during IVF-ET after treatment
Observing the embryo status | through study completion, an average of 1 year
  Observing the grade I embryo ratio, blastocyst formation rate and high quality blastocyst ratio when patients undergoing IVF/ICSI-ET after the treatment
Observing the pregnancy status | through study completion, an average of 1 year
  Observing the biochemical, clinical and ongoing pregnancy rate
Blood corticotropin-releasing hormone (CRH) examination | 0 week and up to 12 weeks
  Observing the level of blood corticotropin-releasing hormone (CRH) at baseline and immediately after treatment
Blood norepinephrine index examination | 0 week and up to 12 weeks
  Observing the level of blood norepinephrine at baseline and immediately after treatment
Blood 5-hydroxytryptamine (5-HT) index examination | 0 week and up to 12 weeks
  Observing the level of blood 5-hydroxytryptamine (5-HT) at baseline and immediately after treatment
Blood beta-aminobutyric acidne (DA) examination | 0 week and up to 12 weeks
  Observing the level of blood beta-aminobutyric acidne (DA) at baseline and immediately after treatment
Blood beta-aminobutyric acid (GABA) examination | 0 week and up to 12 weeks
  Observing the level of blood beta-aminobutyric acid (GABA) at baseline and immediately after treatment
Blood dopamine (DA) examination | 0 week and up to 12 weeks
  Observing the level of blood dopamine (DA) at baseline and immediately after treatment
Blood neuro-endorphin (β-ET) examination | 0 week and up to 12 weeks
  Observing the level of blood neuro-endorphin (β-ET) at baseline and immediately after treatment
Evaluation of anxiety status | 0 week and up to 4 weeks
  Anxiety status will be assessed using Zung anxiety self-rating scale (Zung-SAS) at baseline and immediately after treatment.
Evaluation of depression status | 0 week and up to 4 weeks
  Depression status will be assessed using Zung depression self-rating scale (Zung-SDS) at baseline and immediately after treatment.
Evaluation of quality of life | 0 week and up to 4 weeks
  Quality of life will be assessed by SF-36 at baseline and immediately after treatment..
Evaluation of sleep state | 0 week and up to 4 weeks
  Sleep status will be evaluated using Pittsburgh sleep quality index (PSQI) at baseline and immediately after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hanwang Zhang, Principal Investigator — Huazhong University of Science Tech
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
we use the Clinical Trial Management Public Platform to manage and share our date
Supporting Information: Study Protocol
Time Frame: January, 2027, for 1 year
Access Criteria: only for research